CLINICAL TRIAL: NCT00479830
Title: Health and Cancer Issues in the South Asian Community
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2006-0828
Record Dates: First submitted 2007-05-25; First posted 2007-05-28 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-04

CONDITIONS: Attitude to Health
Keywords: Epidemiology; Health Risks; Questionnaire; Interview; South Asian; Asian Indian; Bangladeshi; Pakistani; Sri Lankan
MeSH Terms: interventions — Focus Groups; Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Group 1: South Asian, Subgroup: Asian Indian, population in the Greater Houston area.
  Interventions: Behavioral: Focus Groups; Behavioral: Questionnaire; Behavioral: Interview
- Group 2: South Asian, Subgroup: Bangladeshi, population in the Greater Houston area.
  Interventions: Behavioral: Focus Groups; Behavioral: Questionnaire; Behavioral: Interview
- Group 3: South Asian, Subgroup: Pakistani, population in the Greater Houston area.
  Interventions: Behavioral: Focus Groups; Behavioral: Questionnaire; Behavioral: Interview
- Group 4: South Asian, Subgroup: Sri Lankan, population in the Greater Houston area.
  Interventions: Behavioral: Focus Groups; Behavioral: Questionnaire; Behavioral: Interview

INTERVENTIONS:
Behavioral: Focus Groups — Eight Focus Groups Consisting of 8-10 Members Each
Behavioral: Questionnaire — To collect data to assess the unmet health and cancer needs of the South Asian population in the Greater Houston area and to determine barriers and other factors that affect health in this population.
Behavioral: Interview — To collect data to assess the unmet health and cancer needs of the South Asian population in the Greater Houston area and to determine barriers and other factors that affect health in this population.

SUMMARY:
The goal of this research study is to learn about the health practices, health knowledge, and attitudes of South Asian Americans who live in Houston or the surrounding area.

DETAILED DESCRIPTION:
If you agree to take part in this study, you will be either be interviewed or participate in a focus group.

For both the interview and the focus group, you will be asked to complete a form that asks questions about your ethnicity, gender, date and place of birth, education level, marital status, native language or language proficiency (your ability to speak different languages), years in the US, and the number of adults and children living in your household. It should take about 10 minutes to complete. You will not be asked to state any of this information aloud in the focus group.

If you are interviewed, you will be asked questions about your personal health and health history, your health practices, including your eating and physical activity habits, health knowledge, and where and how you receive health services and health education.

If you are assigned to a focus group, you will participate in one of 4-8 "focus" (discussion) groups. Each group will have 8-10 participants. A trained focus group moderator will also attend the session, as well as at least 1 member of the research staff. Some groups may have only males. The other groups may have only females.

The moderator may ask you to use your first name with the group. He/she will ask your focus group a series of questions for discussion. As a group, you will be asked to discuss your comments, opinions, and observations. The questions and discussion will relate to your health practices; your knowledge, attitudes, and beliefs about health; your sources of information about health; and any barriers (difficulties) you may have experienced when accessing health care services.

Focus group participants will also be given a draft of a health survey for South Asian Americans that is being developed by researchers. After reading the survey, you will be asked to provide feedback about the cultural relevance and appropriateness of the questions on the survey. In other words, you will discuss whether the questions seem to apply well to the South Asian American community. Researchers are also interested in hearing your feedback about how best to recruit South Asian Americans to complete the health survey.

The interviews will last about 30-40 minutes. Each focus group session will last about 2 hours. The interview and the focus group may be audiotaped so that the participants' responses may be written out and then studied by researchers.

After the interview or focus group session, your participation in this study will be over.

This is an investigational study. Up to 150 individuals will participate in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Self identified South Asian (Asian Indian, Bangladeshi, Pakistani, Sri Lankan) residents of Harris, Fort Bend, Brazoria and Galveston counties.
2. 18 years of age or older
3. Those who speak the languages (including English) that had been identified as most frequently used in Houston's South Asian community by the Community Advisory Committee.

Exclusion Criteria:

1. None
2. Sri Lankans who participated in Protocol 2006-1047.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: South Asian population in the Greater Houston area.
Sampling Method: Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2007-04; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Health Practices, Health Knowledge & Attitudes of South Asian Americans living in Houston | 3+ years
  Data from Interviews + Focus Groups

CONTACTS AND LOCATIONS:
Overall Officials: Richard A. Hajek, PHD, MS, BA, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org